CLINICAL TRIAL: NCT02849067
Title: Hemodynamic Responses of Stable Ischemic Heart Disease Patients to a Comedy Session: Randomized Controlled Trial
Brief Title: Hemodynamic Responses of Stable Ischemic Heart Disease Patients to a Comedy Session
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-0598
Record Dates: First submitted 2016-07-19; First posted 2016-07-29 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Ischaemic Heart Disease
Keywords: ischaemic heart disease; comedy session; laughter therapy
MeSH Terms: conditions — Coronary Artery Disease | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Treatment (Experimental): Patients in this group will watch a comedy show that will will not exceed 30 minutes. This group will have until five patients.
  Interventions: Other: Group Treatment
- Group Control (Other): patients in this group will watch a documentary that will not exceed 30 minutes. This will have until five patients
  Interventions: Other: Group Control

INTERVENTIONS:
Other: Group Treatment — Patients in this group will watch a comedy show that will will not exceed 30 minutes. This group will have until five patients.
  Arms: Group Treatment
Other: Group Control — patients in this group will watch a documentary that will not exceed 30 minutes. This will have until five patients
  Arms: Group Control

SUMMARY:
It is known that laughter can bring benefits in terms of physiological and psychological parameters, in addition to improving the individual's quality of life. However, the literature is still scarce as to the existence of studies investigating the effects of a comedy film specifically in hemodynamics.

DETAILED DESCRIPTION:
Objective: To evaluate the effect of a comedy film session on the cardiac index, Systemic Vascular Resistance and Vascular Resistance Index Systemic in stable ischemic heart disease patients.

Method: Randomized Clinical Trial. Patients will be coming from Ischemic Heart Disease clinic at the Hospital de Clínicas de Porto Alegre (HCPA), all in regular monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 40 and 80 years
* Both female and male
* Diagnosis of ischemic heart disease by cardiac catheterization , with 50% lesion in at least one epicardial vessel

Exclusion Criteria:

* Participants enrolled in another Randomized Clinical trial
* Autoimmune diseases
* Valvulopathy with mechanical or biological cardiac prosthesis
* Presence of pacemakers and implantable cardioverter
* Left bundle branch block in the electrocardiogram (ECG) of 12 derivations
* Severe lung disease
* Depression or Bipolar Disorder
* Atrial Chronic Fibrillation
* Left ventricular dysfunction (ejection fraction <45%)
* Active Infection or neoplasia (not Basal cell carcinoma)
* Chronic Renal Failure
* Illiteracy and inability to understand the consent form

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-05-25 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Cardiography impedance | 28 weeks
  To assess the volumes and fluid passing through the chest at rest and during the exercise session will be used the Cardiography impedance device PhysioFlow, Enduro model (ManatecBiomedical, France).

SECONDARY OUTCOMES:
Humor | 28 weeks
  it will be used the Humor Scale of Brunel

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Stein, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital De Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Polanczyk CA, Ribeiro JP. Coronary artery disease in Brazil: contemporary management and future perspectives. Heart. 2009 Jun;95(11):870-6. doi: 10.1136/hrt.2008.155853. Epub 2009 Mar 3. PMID 19261601
- [Background] Miller M, Mangano C, Park Y, Goel R, Plotnick GD, Vogel RA. Impact of cinematic viewing on endothelial function. Heart. 2006 Feb;92(2):261-2. doi: 10.1136/hrt.2005.061424. No abstract available. PMID 16415199
- [Background] Bennett MP, Lengacher C. Humor and Laughter May Influence Health: II. Complementary Therapies and Humor in a Clinical Population. Evid Based Complement Alternat Med. 2006 Jun;3(2):187-90. doi: 10.1093/ecam/nel014. Epub 2006 Apr 24. PMID 16786047
- [Background] Bennett MP, Lengacher C. Humor and Laughter May Influence Health: III. Laughter and Health Outcomes. Evid Based Complement Alternat Med. 2008 Mar;5(1):37-40. doi: 10.1093/ecam/nem041. PMID 18317546
- [Background] Vlachopoulos C, Xaplanteris P, Alexopoulos N, Aznaouridis K, Vasiliadou C, Baou K, Stefanadi E, Stefanadis C. Divergent effects of laughter and mental stress on arterial stiffness and central hemodynamics. Psychosom Med. 2009 May;71(4):446-53. doi: 10.1097/PSY.0b013e318198dcd4. Epub 2009 Feb 27. PMID 19251872
- [Background] Sugawara J, Tarumi T, Tanaka H. Effect of mirthful laughter on vascular function. Am J Cardiol. 2010 Sep 15;106(6):856-9. doi: 10.1016/j.amjcard.2010.05.011. PMID 20816128
- [Background] Mora-Ripoll R. Potential health benefits of simulated laughter: a narrative review of the literature and recommendations for future research. Complement Ther Med. 2011 Jun;19(3):170-7. doi: 10.1016/j.ctim.2011.05.003. Epub 2011 May 25. PMID 21641524
- [Background] Bennett M, Lengacher C. Use of complementary therapies in a rural cancer population. Oncol Nurs Forum. 1999 Sep;26(8):1287-94. PMID 10497768
- [Background] Lengacher CA, Bennett MP, Kip KE, Keller R, LaVance MS, Smith LS, Cox CE. Frequency of use of complementary and alternative medicine in women with breast cancer. Oncol Nurs Forum. 2002 Nov-Dec;29(10):1445-52. doi: 10.1188/02.ONF.1445-1452. PMID 12432415
- [Background] Miller M, Fry WF. The effect of mirthful laughter on the human cardiovascular system. Med Hypotheses. 2009 Nov;73(5):636-9. doi: 10.1016/j.mehy.2009.02.044. Epub 2009 May 27. PMID 19477604
- [Background] Overeem S, Taal W, Ocal Gezici E, Lammers GJ, Van Dijk JG. Is motor inhibition during laughter due to emotional or respiratory influences? Psychophysiology. 2004 Mar;41(2):254-8. doi: 10.1111/j.1469-8986.2003.00145.x. PMID 15032990
- [Background] Tan SA, Tan LG, Lukman ST, Berk LS. Humor, as an adjunct therapy in cardiac rehabilitation, attenuates catecholamines and myocardial infarction recurrence. Adv Mind Body Med. 2007 Winter;22(3-4):8-12. PMID 20664127
- [Background] Berk LS, Felten DL, Tan SA, Bittman BB, Westengard J. Modulation of neuroimmune parameters during the eustress of humor-associated mirthful laughter. Altern Ther Health Med. 2001 Mar;7(2):62-72, 74-6. PMID 11253418
- [Background] Ishihara S, Nohara R, Makita S, Imai M, Kubo S, Hashimoto T. Immune function and psychological factors in patients with coronary heart disease (I). Jpn Circ J. 1999 Sep;63(9):704-9. doi: 10.1253/jcj.63.704. PMID 10496486
- [Background] LEVI L. THE URINARY OUTPUT OF ADRENALIN AND NORADRENALIN DURING PLEASANT AND UNPLEASANT EMOTIONAL STATES. A PRELIMINARY REPORT. Psychosom Med. 1965 Jan-Feb;27:80-5. doi: 10.1097/00006842-196501000-00009. No abstract available. PMID 14258699
- [Background] Bennett MP, Lengacher CA. Humor and laughter may influence health. I. History and background. Evid Based Complement Alternat Med. 2006 Mar;3(1):61-3. doi: 10.1093/ecam/nek015. Epub 2006 Jan 16. PMID 16550224